CLINICAL TRIAL: NCT03258216
Title: The Traditional Chinese Medicine (TCM) Tongue Diagnosis Indices of Upper Gastrointestinal (UGI) Disorders
Brief Title: TCM Tongue Diagnosis Indices of UGI Disorders
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, hung yu chiang, Director of Chinese Medicine department, Chang Gung Memorial Hospital
Other Study IDs: 104-4725B
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Upper Gastrointestinal Disorders
Keywords: Upper gastrointestinal disorders; Automatic tongue diagnosis system; Panendoscopy
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- peptic ulcer: patients who had upper GI symptoms and diagnosed as peptic ulcer by panendoscopy, followed tongue images by Automatic Tongue Diagnosis System
  Interventions: Diagnostic Test: panendoscopy; Diagnostic Test: tongue image
- healthy: patients who had no past history or systemic disease, diagnosed as UGI negative finding by panendoscopy, followed tongue images by Automatic Tongue Diagnosis System
  Interventions: Diagnostic Test: panendoscopy; Diagnostic Test: tongue image

INTERVENTIONS:
Diagnostic Test: panendoscopy — panendoscopy
Diagnostic Test: tongue image — capture tongue images by Automatic Tongue Diagnosis System

SUMMARY:
The Automatic Tongue Diagnosis System (ATDS) was developed to capture tongue images and extract features reliably to assist the diagnosis of TCM practitioners.This project will employ the ATDS verified to extract the tongue features of patients with upper gastrointestinal disorders, such as peptic ulcer, etc. A TCM indices derived through the non-intrusive tongue diagnosis procedure can provide valuable information for clinical doctors to analyze the current status of a patient and dynamically schedule a treatment plan, facilitating early detection and diagnosis of upper gastrointestinal disorders.

DETAILED DESCRIPTION:
Upper gastrointestinal disorders are common in clinical practice. Currently, the diagnosis of peptic ulcer only depends on laboratory exams such as clinical symptoms, blood test, urine test and feces test. But the result can be only auxiliary exams which don't gain correct diagnosis on helping assess ulcer severity. As the most suitable diagnosis method, panendoscopy can directly observe lesions, judge disease severity, carry out a biopsy, test lesion is benignant or malignant, Helicobacter Pylorus infection or not, the degree of inflammation, etc. But panendoscopy belongs to invasive test. If we can observe tongue characteristics of patients with upper gastrointestinal diseases through scientific tongue diagnosis, physical discomfort caused by the test will be significantly reduced.

Based on clinical observational study, this project will employ the Automatic Tongue Diagnosis System (ATDS) developed. The ATDS was developed to capture tongue images and extract features reliably to assist the diagnosis of TCM practitioners demonstrates the steps in the three major functions, i.e., image capturing and color calibration, tongues area segmentation, and tongue feature extraction, included in the ATDS.

Variations in background lighting may change the color and brightness of the acquired images, greatly affecting consistency and stability of the extracted tongue features. The ATDS developed can automatically correct lighting and color deviation caused by the change of background lighting with a color bar attached in the ATDS. The color bar placed beside the patient is used for color calibration to make sure the image quality is consistent even taken at different circumstances. Tongue images are analyzed by first isolating the tongue region within an image to eliminate irrelevant lower facial portions and background surrounding the tongue, thereby facilitating feature identification and extraction; and then extracting the tongue features by employing criteria such as the aspect ratio, color composition, location, shape, and color distribution of the tongue, as well as the quantity of neighboring pixels. Features including tongue color, tongue fissure, fur color, fur thickness, ecchymosis, tooth mark, red dot, saliva, and tongue shape are extracted to further generate detailed information regarding length, area, moisture, and number of fissures, marks, and dots to be employed in tongue diagnosis. Nine primary tongue features, including tongue color (slightly white, slightly red, red, dark red, dark purple), fur color (white, yellow, dye), fur thickness (none, thin, thick), saliva (none, little, normal, excessive), tongue shape (thin and small, moderate, fat and large), tongue fissure, red dot, ecchymosis, and tooth marks (the last four features are divided into categories of none, mild, moderate, and severe), are selected for tongue diagnosis.

This project will employ the ATDS verified to extract the tongue features of patients with upper gastrointestinal disorders. Through statistically analysis of the data collected and cross-referencing the existing indices of western medicine, we aim to derive meaningful TCM indices from tongue diagnosis of upper gastrointestinal diseases, such as peptic ulcer, etc. A TCM indices derived through the non-intrusive tongue diagnosis procedure can provide valuable information for clinical doctors to analyze the current status of a patient and dynamically schedule a treatment plan, facilitating early detection and diagnosis of upper gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper gastrointestinal disorders
* Both males and females above 20 years old were included
* Patients who had signed Institutional Review Board (IRB) agreement

Exclusion Criteria:

* Patients who had not signed IRB agreement
* Patients who had hypertension, diabetes, hepatitis, or other systemic diseases
* Pregnant women
* Patient with acute infection
* Cognitive impaired, for example, cancer metastasis to brain or dementia
* Risk of temporomandibular joint dislocation
* Patients unable to protrude the tongue stably

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with upper gastrointestinal disorders
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Tongue features | 5-10 mins
  diagnosed by the Automatic Tongue Diagnosis System (ATDS)

SECONDARY OUTCOMES:
Panendoscopy report | 20-30 mins
  diagnosed upper GI disorders by panendoscopy

CONTACTS AND LOCATIONS:
Overall Officials: yu-chiang hung, Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo LC, Cheng TL, Chiang JY, Damdinsuren N. Breast cancer index: a perspective on tongue diagnosis in traditional chinese medicine. J Tradit Complement Med. 2013 Jul;3(3):194-203. doi: 10.4103/2225-4110.114901. PMID 24716178
- [Background] Lo LC, Chiang JY, Cheng TL, Shieh PS. Visual agreement analyses of traditional chinese medicine: a multiple-dimensional scaling approach. Evid Based Complement Alternat Med. 2012;2012:516473. doi: 10.1155/2012/516473. Epub 2012 Sep 17. PMID 23024693
- [Background] Kim J, Son J, Jang S, Nam DH, Han G, Yeo I, Ko SJ, Park JW, Ryu B, Kim J. Availability of tongue diagnosis system for assessing tongue coating thickness in patients with functional dyspepsia. Evid Based Complement Alternat Med. 2013;2013:348272. doi: 10.1155/2013/348272. Epub 2013 Sep 15. PMID 24159343
- [Background] Chiu CC. A novel approach based on computerized image analysis for traditional Chinese medical diagnosis of the tongue. Comput Methods Programs Biomed. 2000 Feb;61(2):77-89. doi: 10.1016/s0169-2607(99)00031-0. PMID 10661393
- [Background] Lee TC, Lo LC, Wu FC. Traditional Chinese Medicine for Metabolic Syndrome via TCM Pattern Differentiation: Tongue Diagnosis for Predictor. Evid Based Complement Alternat Med. 2016;2016:1971295. doi: 10.1155/2016/1971295. Epub 2016 May 25. PMID 27313640
- [Background] Kim J, Han G, Ko SJ, Nam DH, Park JW, Ryu B, Kim J. Tongue diagnosis system for quantitative assessment of tongue coating in patients with functional dyspepsia: a clinical trial. J Ethnopharmacol. 2014 Aug 8;155(1):709-13. doi: 10.1016/j.jep.2014.06.010. Epub 2014 Jun 13. PMID 24933221
- [Background] Lo LC, Chen CY, Chiang JY, Cheng TL, Lin HJ, Chang HH. Tongue diagnosis of traditional Chinese medicine for rheumatoid arthritis. Afr J Tradit Complement Altern Med. 2013 Aug 12;10(5):360-9. doi: 10.4314/ajtcam.v10i5.24. eCollection 2013. PMID 24311851
- [Background] Lo LC, Chen YF, Chen WJ, Cheng TL, Chiang JY. The Study on the Agreement between Automatic Tongue Diagnosis System and Traditional Chinese Medicine Practitioners. Evid Based Complement Alternat Med. 2012;2012:505063. doi: 10.1155/2012/505063. Epub 2012 Aug 8. PMID 22924055
- [Background] Hu J, Han S, Chen Y, Ji Z. Variations of Tongue Coating Microbiota in Patients with Gastric Cancer. Biomed Res Int. 2015;2015:173729. doi: 10.1155/2015/173729. Epub 2015 Sep 17. PMID 26457297
- [Background] Jung CJ, Jeon YJ, Kim JY, Kim KH. Review on the current trends in tongue diagnosis systems. Integr Med Res. 2012 Dec;1(1):13-20. doi: 10.1016/j.imr.2012.09.001. Epub 2012 Oct 5. PMID 28664042
- [Derived] Wu TC, Lu CN, Hu WL, Wu KL, Chiang JY, Sheen JM, Hung YC. Tongue diagnosis indices for gastroesophageal reflux disease: A cross-sectional, case-controlled observational study. Medicine (Baltimore). 2020 Jul 17;99(29):e20471. doi: 10.1097/MD.0000000000020471. PMID 32702810